CLINICAL TRIAL: NCT00482755
Title: A Feasibility Study of Pre-Operative Sunitinib (SU11248) With Multiple Pharmacodynamic Endpoints in Patients With T1c-T3 Operable Carcinoma of the Breast
Brief Title: Sunitinib in Treating Patients With Newly Diagnosed Stage II or Stage III Breast Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA29; CAN-NCIC-MA29 (Other: PDQ Identifier); PFIZER-CAN-NCIC-MA29 (Other: Pfizer); CDR0000547161 (Other: PDQ)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Sunitinib; Immunohistochemistry; Biopsy, Needle; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: sunitinib malate
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: needle biopsy
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with newly diagnosed stage II or stage IIIA breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of neoadjuvant sunitinib malate in patients with newly diagnosed, resectable stage II-IIIA breast cancer.

Secondary

* Determine the nature, severity, and frequency of adverse events in patients treated with this drug.
* Determine the response rate in patients treated with this drug.
* Evaluate markers of angiogenesis (e.g., VEGF receptor, platelet-derived growth factor receptor, circulating plasma VEGF, sVEGFR-2, sVEGFR-3, sKIT, and tumor vascularity) both pre- and post-treatment.
* Examine the role of both host- and tumor-specific genes pertaining to response and toxicity.
* Compare tumor vascular parameters pre- and post-treatment using DCE-MRI.
* Compare cell death and tumor microcirculation pre- and post-treatment using contrast-enhanced spectroscopic and microbubble contrast-enhanced ultrasound.
* Compare tumor metabolic activity pre- and post-treatment using fludeoxyglucose F 18-PET.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily for 14-21 days in the absence of disease progression or unacceptable toxicity.

Tissue samples are obtained by needle biopsy at baseline and once between days 14-21. Blood samples are collected at baseline, once between days 14-21, and at 4 weeks post-treatment for pharmacodynamic and other studies. Markers of angiogenesis (VEGF receptors, platelet-derived growth factor receptor, VEGF, sKIT, and tumor vascularity) are detected by immunohistochemistry. DCE-MRI and fludeoxyglucose F 18-PET are conducted for research studies at baseline and once between days 14-21.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Newly diagnosed disease
  * Stage II-IIIA (T1c, T2, or T3) disease
  * Unifocal disease
  * Resectable disease
* Tumor must be suitable for multiple biopsies and imaging
* No prior breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-1
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine normal
* Calcium ≤ 3 mmol/L
* Bilirubin normal
* ALT and AST ≤ 2.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancies except adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No QTc prolongation (defined as a QTc interval ≥ 500 msec) or other significant ECG abnormalities
* No history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No prior or concurrent NYHA class II-IV cardiovascular disease
* No inadequately controlled hypertension (systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg)
* No myocardial infarction, cardiac arrhythmia, stable or unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within the past 12 months
* No pulmonary embolism within the past 12 months
* No cerebrovascular accident or transient ischemic attack within the past 12 months
* No serious illness or medical condition that would preclude study compliance including, but not limited to, the following:

  * History of significant neurologic or psychiatric disorder
  * Active uncontrolled infection
  * Serious or nonhealing wound, ulcer, or bone fracture
* No medical condition that could interfere with oral medication intake (e.g., frequent vomiting, malabsorption)
* No history of allergic reactions attributed to compounds with similar chemical composition to sunitinib malate
* No preexisting hypothyroidism unless patient is euthyroid on medication

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including the following:

  * Azole antifungals (ketoconazole, miconazole)
  * Verapamil
  * Clarithromycin
  * HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir)
  * Erythromycin
  * Delavirdine
  * Diltiazem
* At least 12 days since prior and no concurrent CYP3A4 inducers, including the following:

  * Rifampin
  * Phenytoin
  * Rifabutin
  * Hypericum perforatum (St. John's wort)
  * Carbamazepine
  * Efavirenz
  * Pentobarbital
  * Tipranavir
  * Phenobarbital
* No prior protein tyrosine kinase inhibitor
* No prior antiangiogenic agent
* No prior hormonal therapy, radiotherapy, chemotherapy, surgery, investigational therapy, or other therapy for breast cancer
* At least 12 days since prior and no concurrent cyclooxygenase-2 inhibitors (e.g., etoricoxib, valdecoxib, celecoxib, dual cyclooxygenase/lipid oxidation, and lumiracoxib)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent agents with proarrhythmic potential (e.g., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide)
* No other concurrent treatment for breast cancer
* No concurrent coumadin-derivative anticoagulants (e.g., warfarin)

  * Anticoagulants at ≤ 2 mg/day for prophylaxis of thrombosis allowed
  * Low molecular weight heparin allowed provided INR ≤ 1.5

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-04-08 (Actual); Primary Completion 2010-03-15 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Feasibility

SECONDARY OUTCOMES:
Nature, severity, and frequency of adverse events
Activity (response rate)
Markers of angiogenesis pre- and post-treatment
Role of both host- and tumor-specific genes pertaining to response and toxicity
Comparison of tumor vascular parameters pre- and post-treatment
Comparison of cell death and tumor microcirculation pre- and post-treatment
Comparison of tumor metabolic activity pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E. Trudeau, BSc, MA, MD, FRCPC, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (2):
- Canada (2):
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No